CLINICAL TRIAL: NCT02832661
Title: BIOMARGIN European, Ambispective Cohort of Adult and Paediatric Renal Transplant Patients for the Evaluation of the Diagnostic and Prognostic Performance of Biomarkers of Renal Graft Injuries
Brief Title: BIOMARGIN European, Ambispective Cohort of Adult and Paediatric Renal Transplant Patients
Acronym: BECS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Collaborators: Hannover Medical School (Other); KU Leuven (Other); Hôpital Necker-Enfants Malades (Other); Hospital Purpan (Other)
Responsible Party: Sponsor
Other Study IDs: I15038; grant agreement no: 305499 (Other Grant/Funding Number: European Community's Seventh Framework Programme (FP7))
Record Dates: First submitted 2015-11-16; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Transplantation
Keywords: renal allograft; graft injuries; biopsy; biomarkers; omics approach

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Urine, plasma, whole blood, biopsy core (only in adults)
Oversight: Data Monitoring Committee: No

SUMMARY:
Biomargin is a European research program aimed at evaluating the diagnostic performance of biomarkers with respect to renal graft injuries, as well as their prognostic performance with respect to 3-year and 5-year graft outcomes.

Nucleic acids, proteins and metabolites previously identified as candidate biomarkers of individual kidney graft lesions will be determined systematically in urine and blood samples collected in patients from the time of transplantation onwards, as well as in the graft tissue when biopsies are required for medical causes or performed systematically in the investigation centres. Their diagnostic and prognostic performance will be checked against histological reading of the biopsies and evolution of the graft function over time.

DETAILED DESCRIPTION:
Background: In renal allograft recipients, 10-year graft survival has not much improved over the past decades. There is thus a need for robust, non-invasive methods to predict and diagnose acute and chronic graft lesions, to improve patient treatment, quality of life and long-term graft survival. Also, there is an unmet need for better understanding of the immune and non-immune mechanisms of interstitial fibrosis /tubular atrophy and graft loss. Several teams have searched for biomarkers of renal graft lesions, but there has been no cross-fecundation of the different "omics" approaches, nor any consolidation of the different clusters of biomarkers discovered using different technologies. An analysis of these different omics levels based on the principles of systems biology is therefore necessary to gain insight into the disease mechanisms and will help to develop predictors at the individual level. Purpose: The European project BIOMARGIN aims to discover, select and validate blood and/or urine biomarkers of renal allograft lesions in adult and paediatric kidney transplant recipients by integrating several omics approaches (mRNA, miRNA, peptides, proteins, lipids and metabolites) in blood, graft tissue and urine. The European cohort study BECS aims to evaluate the diagnostic and prognostic performance of the selected biomarkers over the first 3 and 5 years post-transplantation. Study design: This is a multicenter, international, ambispective, open and non-interventional cohort study, with collection of biological samples. Number of subjects: 450 adult and 50 paediatric renal transplant recipients. Outcomes: The primary endpoint is the graft outcome, assessed at three years as any lesion appeared on graft biopsies after patient enrolment, decline in graft function ≥ 30%, graft loss or patient death. Secondary endpoints include: histological findings in indication biopsies as well as in systematic biopsies (as per centre procedures) at 5 years; cumulated acute rejection episodes; 3-year and 5-year graft survival; and change of renal function assessed by the glomerular filtration rate (GFR) estimated using the MDRD formula. Statistical analysis: The sensitivity, specificity, positive and negative predictive values of the different biomarkers or sets of biomarkers will be evaluated for each of the primary and secondary endpoints. In order to compare the performance of the biomarkers with those of the other known risk factors for the deterioration of renal graft function, longitudinal statistical modelling will be used.

ELIGIBILITY:
Inclusion Criteria for paediatric patients :

* Male or female
* Age between 1 and 17 years inclusive
* Recipient of a kidney allograft in the 24 months prior to enrolment, provided blood and urine samples had been collected between transplantation and enrolment in conditions compatible with those described in this protocol
* Written informed consents of both parents or subject's legally authorized representative prior to any study procedure being performed
* Assent form for the children more than 6 years old

Inclusion Criteria for adult patients:

* Male or female
* Age ≥18 years old (no upper age limit)
* Recipient of a kidney allograft in the 24 months prior to enrolment, provided blood and urine samples had been collected between transplantation and enrolment in conditions compatible with those described in this protocol
* Written informed consent prior to any study procedure being performed

Exclusion Criteria:

* Patients unable to understand the information given by the investigator
* Children less than one year old
* Transplantation of any organ other than the kidney prior or concomitant to the kidney allograft
* Patients returned to dialysis at the time of enrolment

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The eligible patients, 450 adults and 50 pediatrics, will be recruited among the whole list of patients followed for their kidney transplantation in the five investigating centres.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
predictive value of biomarkers | at 3 years post-transplantation

SECONDARY OUTCOMES:
predictive value of biomarkers | at 5 years post-transplantation
Number of biopsy-proven acute rejection episodes | at 1, 3 and 5 years post-transplantation
graft survival at 3 and 5 years post-transplantation | at 3 and 5 years post-transplantation
glomerular filtration rate (GFR in ml/min) estimated using the MDRD formula | over up to 5 years post-transplantation

CONTACTS AND LOCATIONS:
Locations (5):
- University of Leuven - KU Leuven, Leuven, Belgium
- France (3):
  - University Hospital - INSERM, Limoges
  - Necker Children University Hospital, Paris
  - Purpan Children University Hospital, Toulouse
- Medizinische Hochschule Hannover (MHH), Hanover, Germany

REFERENCES:
- [Derived] Vaulet T, Callemeyn J, Lamarthee B, Antoranz A, Debyser T, Koshy P, Anglicheau D, Colpaert J, Gwinner W, Halloran PF, Kuypers D, Tinel C, Van Craenenbroeck A, Van Loon E, Marquet P, Bosisio F, Naesens M. The Clinical Relevance of the Infiltrating Immune Cell Composition in Kidney Transplant Rejection. J Am Soc Nephrol. 2024 Jul 1;35(7):886-900. doi: 10.1681/ASN.0000000000000350. Epub 2024 Apr 19. PMID 38640017
- [Derived] Tinel C, Lamarthee B, Gazut S, Van Loon E, Von Tokarski F, Benon A, Sauvaget V, Garcia-Paredes V, Menager M, Morin L, Aouni L, Cagnard N, Rabant M, Legendre C, Terzi F, Essig M, Gwinner W, Naesens M, Marquet P, Anglicheau D. Modulation of Monocyte Response by MicroRNA-15b/106a/374a During Antibody-mediated Rejection in Kidney Transplantation. Transplantation. 2023 May 1;107(5):1089-1101. doi: 10.1097/TP.0000000000004393. Epub 2023 Apr 22. PMID 36398319
- [Derived] Van Loon E, Gazut S, Yazdani S, Lerut E, de Loor H, Coemans M, Noel LH, Thorrez L, Van Lommel L, Schuit F, Sprangers B, Kuypers D, Essig M, Gwinner W, Anglicheau D, Marquet P, Naesens M. Development and validation of a peripheral blood mRNA assay for the assessment of antibody-mediated kidney allograft rejection: A multicentre, prospective study. EBioMedicine. 2019 Aug;46:463-472. doi: 10.1016/j.ebiom.2019.07.028. Epub 2019 Aug 1. PMID 31378695
- See also: For more information, you can visit the BIOMARGIN website — http://www.biomargin.eu